CLINICAL TRIAL: NCT06169280
Title: A Phase I Study of Repeated Neural Stem Cell-Based Virotherapy and Standard Radiation and Chemotherapy for Newly Diagnosed High-Grade Glioma
Brief Title: Repeated Neural Stem Cell Based Virotherapy for Newly Diagnosed High Grade Glioma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 23C02
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Glioma, Malignant; New Diagnosis Tumor
Keywords: Virotherapy; NSC-CRAd-S-pk7
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Intervention Model Description: Study participants will receive up to 6 doses of NSC-CRAd-S-pk7 in addition to standard of care radiation and temozolomide.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- NSC-CRAd-S-pk7 (Experimental): NSC-CRAd-S-pk7 1·50 x 10⁸ NSCs loaded with1·875 x viral particles administered intra-tumorally on Day 0 and Day 15, then every 4 weeks for up to 6 total doses.
  Interventions: Biological: NSC-CRAd-S-pk7

INTERVENTIONS:
Biological: NSC-CRAd-S-pk7 — NSC-CRAd-S-pk7 1·50 x 10⁸ NSCs loaded with1·875 x viral particles administered intra-tumorally on Day 0 and Day 15, then every 4 weeks for up to 6 total doses.

SUMMARY:
The goal of this clinical trial is to learn about the safety and feasibility of administering repeated doses of neural stem cell (NSC)-conditionally replicative adenovirus (CRAd)-survivin (S)-protomer (p)k7, in persons with newly diagnosed high grade glioma.

The main questions it aims to answer are:

* whether multiple doses of NSC-CRAd-S-pk7 are safe and feasible
* how multiple doses of NSC-CRAd-S-pk7 influence tumor response, overall survival, time to tumor progression, and quality of life.

Participants will:

* undergo a biopsy to confirm high grade glioma, then receive the first dose of NSC-CRAd-S-pk7 into the brain
* about 2 weeks later, undergo surgery to remove the tumor and receive the second dose of NSC-CRAd-S-pk7 into the brain
* start chemoradiation about 2 weeks after surgery, then about 2 weeks later, receive the 3rd dose of NSC-CRAd-S-pk7 into the brain
* four weeks later, at the end of chemoradiation, receive a fourth dose of NSC-CRAd-S-pk7 into the brain.
* after radiation is finished, receive standard of care chemotherapy and tumor-treating fields. Two additional doses of NSC-CRAd-S-pk7 will be given every 4 weeks.

DETAILED DESCRIPTION:
The treatment regimen contains 3 phases:

Surgical phase:

Patients undergo a biopsy and upon intraoperative confirmation of high grade glioma, NSC-CRAd-S-pk7 dose #1 will be injected into the biopsy site. Patients will undergo resection of the tumor 14 (+/- 3) days later, administration of second dose of the investigational product (NSC-CRAd-S-pk7 dose #2), and implantation of the catheter system. The investigational product will then be given monthly for a total of 6 doses (see below).

Radiotherapy phase:

After recovery from surgery (usually within 2 weeks), standard chemoradiotherapy will be initiated consisting of daily radiotherapy (2 Gy per fraction x 30 fractions) and concomitant temozolomide (TMZ) chemotherapy (75 mg/m2 daily from day 1 of RT until last day of RT).

About 10-14 days into radiotherapy (= approx. 4 weeks after intraoperative dose #2), patients will be receiving NSC-CRAd-S-pk7 dose #3 through the previously implanted catheter system. This also marks the beginning of the formal dose-limiting toxicity (DLT) period, as this virus' survivin gene promoter is activated by the concomitant irradiation.

Four weeks later, ie. at the end of radiotherapy dose #4 is administered as previously, provided no DLT toxicity has been observed and viral treatment related toxicities have returned to grade ≤ 2.

Adjuvant (also called maintenance) phase:

As per standard of care, approx. 4 weeks after end of radiotherapy, patients will start maintenance TMZ chemotherapy (150 - 200 mg/m2, daily x 5 every 28 days) and loco-regional treatment with alternating Tumor Treating Fields (TTFields, Optune®). NSC-CRAd-S-pk7 doses #5 and #6 will be administered concurrently (± 3 days) with adjuvant cycle 1 and 2 of TMZ.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a high-grade glioma (WHO grade 3 or grade 4).
* Patients must have presumed high grade glioma (WHO grade 3 or 4) based on clinical and radiologic evaluation for registration.
* A pathologic confirmation of high grade glioma must be made at the time of stereotactic biopsy prior to NSC-CRAd-S-pk7 injection; if this is not possible, the injection will not be performed and the subject will no longer be eligible for the study).
* Tumor must be accessible for injection and must not be located in the brainstem or contained within the ventricular system.
* Planning to undergo standard radiation/chemotherapy.
* 18 years of age or older.
* Performance status (PS) must be WHO PS of < 2.
* Stable or decreasing dose of corticosteroids equivalent to ≤ 6 mg/day for the 5 days prior to inclusion
* Serum glutamic-oxaloacetic transaminase (SGOT or AST) < 3x upper limit of normal
* Serum creatinine < 2mg/dl
* Platelets > 100,000/mm3 and white blood cells (WBCs) > 3000/mm3

Exclusion Criteria:

* Prior or ongoing liver disease including known cirrhosis.
* Known hepatitis B or C infection, known HIV infection.
* Chronic use of immunosuppressive drugs (with exception of corticosteroids required for mass effect).
* Acute viral, bacterial or fungal infections requiring therapy.
* Pregnant or breast-feeding patients.
* Evidence of metastatic disease or other malignancy (except squamous or basal cell skin cancers).
* Prior radiation therapy to the brain or prior treatment for brain tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity of repeat NSC-CRAd-S-pk7 dosing | 8 weeks
  Determination of the dose limiting toxicity of repeated dosing of NSC-CRAd-S-pk7

SECONDARY OUTCOMES:
Objective response to therapy | 5 years
  Objective response to therapy as determined by Immune Response Assessment in Neuro-Oncology (iRANO) criteria
Overall survival | 5 years
  Overall survival time from the first study product injection to death
Progression-free survival | 18 months
  Time from the first study product injection to first confirmed disease progression as determined by objective tumor response

OTHER OUTCOMES:
Functional Assessment of Cancer Therapy-Brain (FACT-Br) score change | 22 weeks
  Change in score on FACT-Br over time as a measure of quality of life, with scores ranging from 0-200; higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Stupp, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared with other researchers.

REFERENCES:
- [Background] Ahmed AU, Thaci B, Tobias AL, Auffinger B, Zhang L, Cheng Y, Kim CK, Yunis C, Han Y, Alexiades NG, Fan X, Aboody KS, Lesniak MS. A preclinical evaluation of neural stem cell-based cell carrier for targeted antiglioma oncolytic virotherapy. J Natl Cancer Inst. 2013 Jul 3;105(13):968-77. doi: 10.1093/jnci/djt141. PMID 23821758
- [Background] Ahmed AU, Thaci B, Alexiades NG, Han Y, Qian S, Liu F, Balyasnikova IV, Ulasov IY, Aboody KS, Lesniak MS. Neural stem cell-based cell carriers enhance therapeutic efficacy of an oncolytic adenovirus in an orthotopic mouse model of human glioblastoma. Mol Ther. 2011 Sep;19(9):1714-26. doi: 10.1038/mt.2011.100. Epub 2011 May 31. PMID 21629227
- [Background] Fares J, Ahmed AU, Ulasov IV, Sonabend AM, Miska J, Lee-Chang C, Balyasnikova IV, Chandler JP, Portnow J, Tate MC, Kumthekar P, Lukas RV, Grimm SA, Adams AK, Hebert CD, Strong TV, Amidei C, Arrieta VA, Zannikou M, Horbinski C, Zhang H, Burdett KB, Curiel DT, Sachdev S, Aboody KS, Stupp R, Lesniak MS. Neural stem cell delivery of an oncolytic adenovirus in newly diagnosed malignant glioma: a first-in-human, phase 1, dose-escalation trial. Lancet Oncol. 2021 Aug;22(8):1103-1114. doi: 10.1016/S1470-2045(21)00245-X. Epub 2021 Jun 29. PMID 34214495
- [Background] Kim CK, Ahmed AU, Auffinger B, Ulasov IV, Tobias AL, Moon KS, Lesniak MS. N-acetylcysteine amide augments the therapeutic effect of neural stem cell-based antiglioma oncolytic virotherapy. Mol Ther. 2013 Nov;21(11):2063-73. doi: 10.1038/mt.2013.179. Epub 2013 Jul 25. PMID 23883863
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009